CLINICAL TRIAL: NCT04052477
Title: Social Web Mining for Suicide Prevention of Young People
Brief Title: Social Web Mining for Suicide Prevention
Acronym: Don't Do It
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: LIRMM - Montpellier - France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0320
Record Dates: First submitted 2019-07-12; First posted 2019-08-09 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Suicidal Behaviors
Keywords: Suicide; Prevention; Social network
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to a recent and alarming WHO (World Health Organisation) report (September 4, 2014), one person dies of suicide every 40 seconds in the world. Suicide is the third-leading cause of death for 15- to 24-year-olds, according to the Centers for Disease Control and Prevention , after accidents and homicide.

This major public health issue need prevention strategies especially directed to at-risk populations. Since 2013, more than 2 billion users are enrolled in social networks such as Twitter or Facebook. Young adults (ages 18 to 29) are the most likely to use social media - fully 90% do.

Consequently, in this project, we focus on suicide prevention in social media network..

The aim of this project is the validation of the algorithm. This algorithm build a decision support system that monitor young people at-risk based on large volume of heterogeneous data collected through social media to improve suicide prevention.

DETAILED DESCRIPTION:
This study is composed of two steps :

1. 9 subjects were recruited. After patients agreement, computer scientists were accessing to patient social network profile. Computer scientists were not able to visualize the content of publications, just run the algorithm that will analyse the content of messages (text, frequency, emoticons…)

   The algorithm defines the 3 most at-risk periods of suicide behaviors, on the next month. This result were compared to periods found by psychiatric interview. The psychiatrist then confirmed or not to LIRM whether periods found by the algorithm conrrespond to those defined by the psychitrist. No data of the social network were collected.
2. the 2nd step aim to improve the algorithm by collecting sociodemographic and clincal data related to patients included.

ELIGIBILITY:
Inclusion criteria:

* Major patient
* Minor patient with parents approval
* Patient hospitalized due to suicide attempt or suicide ideations
* Frequent active user of social netword (Facebook, Instagram, Youtube, Twitter)

Exclusion criteria:

- Patient's refusal to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (major or minor) presenting suicidal behaviors (recent suicide attempt or suicidal ideations)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
sensitivity of the algorithm | 1 day
  baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Guillaume, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC